CLINICAL TRIAL: NCT06019689
Title: Exploratory Study of a Culturally Adapted Manual-assisted Problem-solving Mobile Based Intervention (CAMI) for Suicidal Ideation: A Multicentre, Two Arm, Randomized Controlled Trial From Pakistan
Brief Title: Culturally Adapted Manual-assisted Problem Solving Training Based Mobile Intervention
Acronym: CAMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PILL-CAMI
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Suicidal Ideation
Keywords: self-harm; suicidal ideation; Mobile intervention; cultural adaptation; Pakistan; LMIC; Problem-solving; CBT
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: multicenter exploratory RCT
Who Masked: Outcomes Assessor
Masking Description: Researcher conducting assessments will be masked to participant group allocation. This will be achieved by briefing participants and research staff in advance around maintaining masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Digitally delivered CMAP intervention through App. CMAP is a manual-assisted intervention which has been adapted from a self-help guide called Life After Self-Harm based on the principles of Cognitive behavioral therapy (CBT).
  Interventions: Behavioral: CAMI
- Standard Routine Care (No Intervention): Local medical, psychiatric and primary care services providing standard routine care to participant patients. Participants receiving an initial assessment along with TAU as ascertained by their treating doctor at the hospital or their primary care physician (general practitioner (GP)

INTERVENTIONS:
Behavioral: CAMI — Culturally Adapted manual-assisted problem solving training based Mobile Intervention (CAMI) for Suicidal Ideation. CMAP is a manual-assisted intervention which has been adapted from a self-help guide called Life After Self-Harm based on the principles of Cognitive behavioral therapy (CBT). This intervention is an evaluation of suicidal ideation, crisis skills, problem-solving and CBT techniques to manage emotions, negative thinking, interpersonal relationships and relapse prevention strategies.
  Arms: Intervention

SUMMARY:
Determine the feasibility, acceptability and efficacy of an adapted digitally delivered CMAP (CMAP-SI) intervention (CAMI) compared to treatment as usual (TAU) for patients presenting with suicidal ideation.

DETAILED DESCRIPTION:
The reported suicide rates in South Asia are high compared to the global average. These figures are likely to be an underestimate since suicide data from many LMICs such as Pakistan is lacking and what is available is not reliable (Jordans et al., 2014). According to an estimate, 5,000 to 7,000 suicides take place each year in Pakistan (Hafeez, 2016) and at least 10 to 20 suicide attempts happen for every suicide.

Mobile health is a novel and emerging field in psychiatric and psychological care and treatment of mental health difficulties, it involves the use of telecommunications to provide health care, support and intervention from a distance.

The proposed study will be carried out in two phases; Stage 1) adaptation of an already existing culturally adapted manual assisted problem solving intervention (CMAP) for patients with suicidal ideation presenting to primary care in Pakistan and further adaptation into a digital intervention.

Stage 2) feasibility Randomised Control trial.

ELIGIBILITY:
Inclusion Criteria:

Individuals (aged 18-64) screened and identified as having suicidal ideation

* Able to give written informed consent
* Living within the catchment areas of participating hospitals
* Have a smart phone and able to operate it
* Able to read and speak Urdu
* Not requiring in-patient psychiatric treatment.

Exclusion Criteria:

* Presence of a diagnosed physical or intellectual disability as it can prevent individuals from engaging with the intervention. This will be assessed by the research team at screening stage. Any disabilities will be identified by a relevant clinician (e.g. Psychiatrist).
* Temporary resident unlikely to be available for follow-up (b) participants with a diagnosis of DSM-IV mental disorder due to general medical condition or substance misuse, dementia, delirium, alcohol and drug dependence, schizophrenia, or bipolar disorder.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicide Ideation . | Change in scores from baseline to 3 and 6-month post-randomization
  The BSI is a 19-item self-report instrument for detecting and measuring the current intensity of the patient's attitudes, behaviors and specificity of a patient's thoughts to die by suicide during the past week. Higher scores indicate greater severity of suicidal ideation

SECONDARY OUTCOMES:
Depression | Change in scores from baseline to 3 and 6-month post-randomization
  Beck Depression Inventory (BDI), which is a 21-item scale measuring symptoms of depression. Higher scores on the scale indicate greater severity of depression.
Hopelessness | Change in scores from baseline to 3 and 6-month post-randomization
  Beck Hopelessness Scale (BHS) (Beck, A and Steer, R, 1988) is a self-report instrument designed to measure three aspects of hopelessness: feelings about the future, loss of motivation and expectations during the past week. Higher scores indicate greater severity of hopelessness.
Health-related quality of life | Change in scores from baseline to 3 and 6-month post-randomization
  Quality of life-EuroQoL (EQ-5D) (Brooks, R. and Group, E., 1996): This is a standardised instrument to measure health-related quality of life. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Higher scores indicate better quality of life.
Client Service Receipt Inventory | Change in scores from baseline to 3 and 6-month post-randomization
  Detailed description of the use of health services will be collected using the Client Service Receipt Inventory (CSRI)
Client Satisfaction Questionnaire | level of satisfaction at end of intervention i.e., 3-month post-randomization
  The Client Satisfaction Questionnaire (Attkisson, Zwick, & planning, 1982) is an 8 item measure of client satisfaction with services. Higher scores indicate greater satisfaction with the services received.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MRC Psych, FRC Psych, Principal Investigator — Pakistan Institute of Living and Learning
Locations (7):
- Pakistan (7):
  - Quetta Site, Quetta, Balochistan
  - Peshawar Site, Peshawar, KPK
  - Lahore Site, Lahore, Punjab Province
  - Multan Site, Multan, Punjab Province
  - Rawalpindi Site, Rawalpindi, Punjab Province
  - Hyderabad Site, Hyderābād, Sindh
  - Karachi Site, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husain N, Kiran T, Chaudhry IB, Williams C, Emsley R, Arshad U, Ansari MA, Bassett P, Bee P, Bhatia MR, Chew-Graham C, Husain MO, Irfan M, Khaliq A, Minhas FA, Naeem F, Naqvi H, Nizami AT, Noureen A, Panagioti M, Rasool G, Saeed S, Bukhari SQ, Tofique S, Zadeh ZF, Zafar SN, Chaudhry N. A culturally adapted manual-assisted problem-solving intervention (CMAP) for adults with a history of self-harm: a multi-centre randomised controlled trial. BMC Med. 2023 Jul 31;21(1):282. doi: 10.1186/s12916-023-02983-8. PMID 37525207